CLINICAL TRIAL: NCT06194396
Title: Effect of Chlorhexidine 2% Versus Alcohol on Healthcare Associated Infections in Neonates: Randomized Control Trial
Brief Title: Effect of Chlorhexidine Versus Alcohol on Infections in Neonates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Ali El-Farrash, Principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU
Record Dates: First submitted 2023-05-04; First posted 2024-01-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Neonatal Infection
MeSH Terms: interventions — Chlorhexidine; Ethanol

STUDY DESIGN:
Intervention Model Description: 2 groups 50 neonates / group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50 neonates using alcohol (Active Comparator): Alcohol will be used as skin disinfectant before insertion of the central venous catheter, PICC line, and umbilical venous catheter and during its routine care
  Interventions: Other: alcohol
- 50 neonates using chlorhexidine (Experimental): Chlorhexidine will be used as skin disinfectant prior to insertion of the central venous catheter, PICC line, and umbilical venous catheter and during its routine care
  Interventions: Other: chlorhexidine

INTERVENTIONS:
Other: chlorhexidine — chlorhexidine will be used as skin disinfectant before insertion of CVC, PICC line, and umbilical catheter
  Arms: 50 neonates using chlorhexidine
Other: alcohol — alcohol will be used as skin disinfectant before insertion of CVC ,PICC line and umbilical catheter
  Arms: 50 neonates using alcohol

SUMMARY:
Chlorhexidine is a local antiseptic that has an important role in the prevention of catheter-associated bloodstream infections. Its application to a newborn's umbilical cord reduces all-cause neonatal mortality.

DETAILED DESCRIPTION:
Skin disinfection by an appropriate antiseptic agent is essential to prevent healthcare-associated infection. Common pathogens responsible for sepsis have been detected in skin microbiota of hospitalized neonates. Such skin inhabitants can cause sepsis and also lead to blood culture contamination resulting in unnecessary antibiotic use. Strict asepsis bundles have been shown to reduce catheter-related blood stream infection (CRBSI) and contamination rates. The choice of appropriate skin disinfectant is, however, based on low-quality evidence, even in adults.

Chlorhexidine gluconate (CHG) is a broad-spectrum antiseptic which is effective against a host of neonatal pathogens. CHG-based products are used frequently in the healthcare setting for peripheral and central venous catheter (CVC) site skin preparation, daily bathing of intensive care unit patients, full-body newborn skin cleansing, umbilical cord care, and Staphylococcus aureus decolonization.

In neonates, CHG used as antiseptic for CVC insertion site preparation and maintenance decreases CVC tip microbial colonization. Trials of full-body skin cleansing and umbilical cord care with CHG in the developing world, which included infants less than 34 weeks gestational age, have demonstrated reduced risk of neonatal mortality. Despite proven efficacy of CHG in neonates, current guidelines acknowledge that no recommendations with regards to CHG antisepsis can be made for infants less than 2 months of age due to incomplete safety data in this population.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with gestational age 28 weeks or more.
* Neonates needing the insertion of a peripherally inserted central catheter (PICC line) or CVC or umbilical catheter.

Exclusion Criteria:

* Extremely preterm (GA less than 28 weeks).
* Babies who have an allergy to chlorhexidine 2%.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
reduction in health care acquired neonatal infection | 8 months
  to determine whether the use of chlorhexidine 2% solution reduces the health care-acquired neonatal infection when compared to alcohol

CONTACTS AND LOCATIONS:
Overall Officials: Rania El Farrash, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No